CLINICAL TRIAL: NCT06900634
Title: Utilizing Implementation Research Methodologies to Adapt an Intervention to Reduce Alcohol Use and Improve HIV Care Outcomes Among Men Living With HIV Who Have Serodiscordant Pregnant Partners
Brief Title: Pilot of an Intervention to Reduce Alcohol Use and Improve ART Adherence Among Men Living With HIV With Pregnant Partners in Uganda.
Acronym: Kisoboka Amaka
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-2024-0098; K01AA031208 (NIH)
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: HIV Antiretroviral Therapy (ART) Adherence; Alcohol Consumption
Keywords: hiv; motivational interviewing; behavioral economics; alcohol use disorder
MeSH Terms: conditions — Alcohol Drinking; Acquired Immunodeficiency Syndrome; Alcoholism | interventions — Mass Screening; Referral and Consultation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kisoboka Amaka (Experimental)
  Interventions: Behavioral: Kisoboka Amaka
- Screening and Referral (Active Comparator)
  Interventions: Behavioral: Screening and Referral

INTERVENTIONS:
Behavioral: Kisoboka Amaka — KISOBOKA AMAKA intervention adapts and combines a behavioral intervention with a structural component. The behavioral intervention component includes, alcohol screening, financial literacy training, and counseling and goal setting related to savings, alcohol use, and HIV care engagement. The structural intervention component focuses on depositing earnings into mobile savings programs. Kisoboka Amaka content will be "finalized" in aims 1 and 2. However, we expect core intervention components to remain unchanged including: 4 counseling sessions (2 individual, 2 group), 2x weekly text message reminders of goals and mobile money set up. Potential additional components include: 1 family focused couples session, self monitoring of alcohol use (via mobile breathalyzer) and PEth (an objective biomarker measure of alcohol use) boosted alcohol counseling.
  Arms: Kisoboka Amaka
Behavioral: Screening and Referral — Alcohol screening and referral and emphasizing the importance of HIV care engagement and ART adherence
  Arms: Screening and Referral

SUMMARY:
Hazardous alcohol use, which is common among men in Uganda, is a primary driver of both HIV risk and intimate partner violence (IPV) in this setting. Among men living with HIV, alcohol use is associated with non-adherence to antiretroviral therapy (ART) and a detectable viral load, increasing the risk of onward HIV transmission to partners. This risk is further heightened when the partner is pregnant, due to the potential for vertical transmission. Therefore, addressing factors that interfere with optimal HIV care outcomes among men living with HIV is critical to HIV prevention in pregnant women.

The goal of this randomized controlled trial (RCT) is to pilot test an intervention that combines alcohol reduction and economic strengthening to improve ART adherence. The study will assess implementation outcomes and preliminary efficacy among men living with HIV who engage in hazardous alcohol use and their pregnant partners (n=30 couples). The main questions it aims to answer are:

1. What are the implementation outcomes (acceptability, appropriateness, feasibility, fidelity, and safety) at the individual, implementer, and organizational levels, and what bridging factors may impede success (e.g., community-academic partnership)?
2. Does the intervention reduce hazardous alcohol use and improve ART adherence among men living with HIV?

Researchers will compare the intervention group (n=15 couples) to the standard of care group (n=15 couples) to determine if the intervention leads to behavior change in alcohol use and ART adherence among men living with HIV.

Participants will:

1. Men in the intervention group will receive the Amaka intervention, designed to reduce alcohol use and improve ART adherence.
2. Complete assessments on hazardous alcohol use, ART adherence, and implementation outcomes at multiple time points (baseline, 3 and 6 months).
3. Engage with implementers to provide post-implementation feedback on feasibility and acceptability.

DETAILED DESCRIPTION:
Men in Uganda who drink heavily face serious health and social challenges, including difficulty staying on HIV treatment, which increases the risk of passing HIV to their partners. Pregnant women in serodiscordant relationships, where the male partner has HIV but the woman does not, are at especially high risk of infection. Reducing alcohol use and improving HIV treatment adherence in men is critical to protecting both their partners and future children from HIV.

To address this issue, researchers previously developed Kisoboka ("It is possible"), an intervention designed to help men reduce alcohol use and engage in HIV care. The original Kisoboka program, tested among fisherfolk in Uganda, combined counseling, text message reminders, and economic strengthening-helping participants open and save money in mobile banking accounts-to improve long-term financial planning while reducing alcohol-related harm. The study found that Kisoboka successfully helped men reduce alcohol use and improve HIV care, but many participants continued drinking at risky levels, suggesting the need for additional support.

The present study adapts Kisoboka for a new population: men living with HIV who are not part of fishing communities but have pregnant partners who do not have HIV. The adapted version, called Kisoboka Amaka ("It is possible, Family!"), maintains the core elements of the original intervention while introducing new strategies tailored to this population, including couples' communication support and biofeedback on alcohol use using biomarker testing or mobile phone breathalyzers.

To ensure the program meets the needs of this new group, the study will first gather input from men living with HIV, their pregnant partners, and healthcare providers to identify necessary modifications (AIM 1). Researchers will explore whether adding biofeedback tools, such as alcohol biomarker tests or mobile phone breathalyzers, could enhance counseling by giving participants a clearer picture of their alcohol use. They will also assess whether a couples' session could improve communication and shared financial goal-setting.

Once these insights are gathered, the intervention will be refined through a collaborative process that includes community members, healthcare providers, and policymakers (AIM 2). Participants will review intervention materials in a process known as theater testing, where they can provide feedback before final adjustments are made. This step ensures that the intervention is both culturally relevant and practically feasible.

Finally, the adapted Kisoboka Amaka program will be tested in a small randomized controlled trial (AIM 3). Thirty couples will be randomly assigned to either receive the intervention or standard care. The study will assess whether Kisoboka Amaka is acceptable and feasible for both participants and providers and will gather preliminary evidence on its potential to reduce hazardous alcohol use and improve adherence to HIV treatment.

By adapting a proven intervention rather than developing a new one from scratch, this study builds on existing evidence while tailoring the program to meet the needs of a different at-risk group. If successful, Kisoboka Amaka could be scaled up to improve HIV prevention and family health across Uganda, helping protect more women and children from HIV while supporting men in reducing alcohol use and staying engaged in HIV care.

ELIGIBILITY:
Inclusion Criteria:

FOR MEN

1. living with HIV;
2. AUDIT-C positive (≥4) indicating potential hazardous drinking;
3. >6 months since initial antiretroviral treatment (ART) initiation;
4. an indicator of potential suboptimal treatment as prevention (TasP) either: (i) last HIV viral load test (within 6 months) was detectable (>20) or (ii) last viral load test between 6 and 13 months ago was detectable (>20) and reports missing ≥2 ART doses in the past 2 weeks or (iii) a lack of viral load test results for the prior 13 months in clinic records and reports missing ≥2 ART doses in the past 2 weeks
5. not planning to move from the area within the next 6 months;
6. have their own mobile phone and can be reached via phone.

FOR WOMEN

1. 18+ years of age (or emancipated minor)
2. Pregnant
3. HIV negative

FOR COUPLES (IF INDIVIDUAL ELIGIBILITY CRITERIA ABOVE ARE MET)

1. married/living together >6 months;
2. planning to stay together >6 months
3. lived in the area for >3 months and
4. not planning to move within <6 months.
5. similar responses on Couple Verification Screening (CVS) form, an instrument to determine if couples are legitimate (e.g., asking each person what they ate the last time they shared a meal with their partner).

Exclusion Criteria:

FOR MEN

1. visibly intoxicated at enrollment (eligible to enroll when not intoxicated);
2. does not speak Luganda or English;
3. currently receiving a majority of work payments via mobile money/digital payments;
4. participated in the Kisoboka pilot RCT;
5. unable to read basic Luganda or English

FOR WOMEN For safety purposes, we will not enroll women who do not feel they can safely participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2027-02-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Antiretroviral therapy adherence | measured at baseline, 3 and 6 months follow up
  ART adherence, measured by level of ARVs detected via blood sample (DBS). Complete adherence (100%) will be defined as TDF >1250 fmol/punch, 700-1249 fmol/punch indicates 4-6 doses per week, 350-699 fmol/punch indicates 2-3 doses per week and <350 fmol/punch indicates <2 doses per week.
Alcohol reduction (change in PEth) | measured at baseline and 6 months follow up
  Reduction in PEth (Non-heavy use will be defined as a PEth result ≥20 ng/ml but <200 ng/ml156. Chronic/heavy use via PEth will be defined as a PEth result ≥200 ng/ml156.*this high threshold was selected due to high levels of heavy alcohol use among MLWH in Uganda).

SECONDARY OUTCOMES:
Alcohol reduction (self report) | measured at baseline 3 and 6 months follow up
  Self-reported hazardous use (AUDIT-C >3).

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University Walter Reed Program, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data from Aims 1 and 2 will be used to develop, theater test, and pilot an intervention and will not generate generalizable knowledge; thus, they are not subject to the NIH Data Sharing Policy. However, data from the Aim 3 pilot study-including raw questionnaire and biological specimen data-will be shared via the NIAAADA repository. All data will be de-identified, with global unique identifiers assigned through the NIMH NDA. Identifiable information will be stored separately and securely for future contact but will not be shared. Survey datasets will be preserved and made available upon request. Audio files and verbatim transcripts from Aim 3 qualitative work will not be shared due to the high risk of participant identification given the purposive sampling and limited geographic area. Instead, we will share codes derived from the qualitative transcripts with NIAAADA.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will not have data for sharing in the first three years of the study and will delay our first submission by updating submission dates (per the NIAAADA guidance). The research community will gain access to the uploaded data when the award ends. As required by NIAAADA, we will also create studies that contain the data used for every publication (except in instances where this data doesn't meet NIH sharing requirements, as described under #2) and include the digital object identifiers (DOI) for that study in the manuscript to aid in findability. NIAAADA will make decisions about how long to preserve the data.
Access Criteria: Data will be findable for the research community through the NIMH Data Archive (NIAAA Data Archive specifically) which is established at the time of study funding. For all publications, an NIAAA Data Archive study will be created. Each of those studies is assigned a digital object identifier (DOI). This data DOI will be referenced in the publication. Investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NIAAA Data Archive repository data by submitting a data access request in accordance with applicable NIAAA Data Archive repository policies. Data requests will be reviewed and granted by an NIMH/NIAAA Data Archive Data Access Committee.
URL: https://nda.nih.gov/nda/access-data-info